CLINICAL TRIAL: NCT07290751
Title: Intravenous Thrombolysis Combined With Tirofiban in Acute Ischemic Stroke: A Multicenter, Prospective, Double-Blind, Placebo-Controlled, Randomized Controlled Trial
Brief Title: Intravenous Thrombolysis Combined With Tirofiban in Acute Ischemic Stroke
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaochuan Huo, Director, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-013
Record Dates: First submitted 2025-08-29; First posted 2025-12-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; tirofiban; thrombolysis
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Tirofiban; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - Tirofiban (Experimental)
  Interventions: Drug: Tirofiban
- Arm B - Placebo (Placebo Comparator)
  Interventions: Other: Placebo (0.9% normal saline)

INTERVENTIONS:
Drug: Tirofiban — After intravenous thrombolysis, if neurological improvement is insufficient (NIHSS score decrease <2 within 1 hour or NIHSS increase ≥1), tirofiban infusion is initiated within 1 hour. The regimen consists of 0.4 μg/kg/min for 30 minutes, followed by 0.1 μg/kg/min for 23.5 hours (total 24 hours). At the 20th hour of infusion, oral antiplatelet therapy (aspirin 100 mg once daily and/or clopidogrel 75 mg once daily) is initiated, overlapping with tirofiban for 4 hours (bridge therapy). At 24 hours, tirofiban infusion is completed, and patients continue oral antiplatelet therapy per protocol.
  Arms: Arm A - Tirofiban
Other: Placebo (0.9% normal saline) — Matched normal saline infusion using the same dosing schedule and pump rates as the tirofiban arm (0.4 μg/kg/min for 30 minutes, then 0.1 μg/kg/min for 23.5 hours; total 24 hours). At the 20th hour of infusion, oral antiplatelet therapy (aspirin 100 mg once daily and/or clopidogrel 75 mg once daily) is initiated, overlapping with placebo infusion for 4 hours (bridge therapy). At 24 hours, placebo infusion is completed, and patients continue oral antiplatelet therapy per protocol.
  Arms: Arm B - Placebo

SUMMARY:
This multicenter, prospective, double-blind, placebo-controlled, randomized trial (ANGEL-DRUG2) aims to evaluate the efficacy and safety of intravenous tirofiban following intravenous thrombolysis in patients with acute ischemic stroke who show insufficient neurological improvement after initial treatment. Eligible patients (≥18 years, baseline NIHSS ≥4, within 4.5 hours from last known well) will be randomized 1:1 to receive either tirofiban or placebo infusion for 24 hours, followed by standard oral antiplatelet therapy. The primary endpoint is the proportion of patients achieving functional independence (mRS 0-2) at 90 days. Secondary outcomes include changes in NIHSS score, vessel recanalization, infarct volume, distribution of mRS scores, recurrent stroke, and health-related quality of life. Safety outcomes focus on symptomatic intracranial hemorrhage and all-cause mortality. Approximately 976 patients will be enrolled across 30 sites in China.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is a leading cause of death and disability worldwide. Intravenous thrombolysis (IVT) and endovascular therapy (EVT) are guideline-recommended treatments, but many patients continue to experience unsatisfactory neurological recovery after IVT alone. Early antiplatelet therapy is recommended as adjunctive management, and tirofiban, a selective and reversible intravenous glycoprotein IIb/IIIa receptor inhibitor, has shown promise in reducing platelet aggregation and thrombus formation without significantly increasing symptomatic intracranial hemorrhage. However, robust evidence regarding its efficacy and safety in AIS patients with poor neurological improvement after IVT is lacking.

ANGEL-DRUG2 is designed to fill this knowledge gap. This trial will enroll 976 patients at 30 centers who present with acute ischemic stroke, have received IVT within 4.5 hours of onset, and demonstrate poor or worsening neurological improvement within 1 hour post-IVT (defined as NIHSS score decrease <2 or increase ≥1). Patients will be randomized in a 1:1 ratio, stratified by center, to receive either tirofiban infusion (0.4 μg/kg/min for 30 minutes, then 0.1 μg/kg/min for 23.5 hours) or placebo (normal saline) infusion of the same regimen. Both groups will be transitioned at 20 hours to standard oral antiplatelet therapy (aspirin and/or clopidogrel).

The primary efficacy endpoint is the proportion of patients achieving a modified Rankin Scale (mRS) score of 0-2 at 90±7 days. Secondary efficacy endpoints include NIHSS change at 36±12 hours, vessel recanalization on CTA/MRA, infarct volume, distribution of mRS scores at multiple timepoints, recurrent stroke within 90 days, and EQ-5D-5L quality-of-life scores. Safety endpoints include symptomatic intracranial hemorrhage within 48 hours (Heidelberg criteria), any intracranial hemorrhage, and all-cause mortality at 90 days.

This rigorously designed study will provide high-quality evidence regarding whether tirofiban, when added to IVT in AIS patients with poor early response, can improve functional outcomes without unacceptable safety risks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Pre-stroke modified Rankin Scale (mRS) score of 0-1.
3. Acute ischemic stroke symptoms within 4.5 hours of last known well time.
4. Baseline National Institutes of Health Stroke Scale (NIHSS) score ≥4.
5. Poor neurological improvement 1 hour after intravenous thrombolysis, defined as NIHSS decrease <2 points, or neurological worsening within 1 hour, defined as NIHSS increase ≥1 point.
6. Not planned for or not eligible for endovascular treatment.
7. Subject or legally authorized representative can provide written informed consent.

Exclusion Criteria:

1. Evidence of intracranial hemorrhage on imaging before randomization.
2. Non-ischemic intracranial pathologies, such as vascular malformation, aneurysm, tumor, abscess, or demyelinating disease.
3. Large or medium vessel stenosis requiring thrombectomy or intra-arterial thrombolysis.
4. Contraindications to tirofiban, including but not limited to:Known hypersensitivity to tirofiban; Severe hepatic dysfunction (ALT >2× ULN or AST >2× ULN); Severe renal dysfunction (serum creatinine >1.5× ULN); Advanced heart failure (NYHA class III-IV); Coagulation disorders or history of systemic bleeding; History of thrombocytopenia or neutropenia; Prior drug-induced hematologic disease or liver dysfunction; Leukopenia (<2×10^9/L) or platelet count <100×10^9/L.
5. Use of tirofiban or other GP IIb/IIIa inhibitors before randomization, or planned use of such agents after randomization.
6. Definite cardioembolic source, including but not limited to: chronic or paroxysmal atrial fibrillation, sick sinus syndrome, mitral stenosis, mechanical prosthetic heart valves, infective endocarditis, history of intracardiac thrombus, myocardial infarction within 3 months, dilated cardiomyopathy, spontaneous left atrial echo contrast, or left ventricular ejection fraction <30%.
7. Pregnancy or lactation.
8. Expected survival <6 months.
9. Pre-existing neurological or psychiatric disorders that may interfere with outcome assessment.
10. Unlikely to complete 90-day follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with mRS 0-2 at 90 days | 90±7 days post-randomization
  Proportion of patients with Modified Rankin Scale (mRS) 0-2, Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.
Symptomatic Intracranial Hemorrhage (sICH) within 48 hours | Randomization to 48 hours
  Heidelberg Bleeding Classification with clinical worsening criteria.

SECONDARY OUTCOMES:
Change in NIHSS from baseline to 36±12 hours | 36±12 hours post-randomization
  Change in National Institute of Health stroke scale score from baseline.The NIH Stroke Scale (NIHSS) score ranges from 0 to 42 points, with lower scores indicating better neurological function
Vascular recanalization rate assessed by CT/MR angiography | 36±12 hours post-randomization
  Vascular recanalization rate assessed by CT/MR angiography
Change in infarct volume at 7±3 days/discharge | 7±3 days post-randomization or discharge
  Change in infarct volume
mRS distribution | 7±3 days/discharge；90±7 days post-randomization
  Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.
Proportion with mRS 0-1 at 90 days | 90±7 days
  Proportion of patients with Modified Rankin Scale (mRS) 0-1, Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.
Proportion with mRS 0-3 at 90 days | 90±7 days
  Proportion of patients with Modified Rankin Scale (mRS) 0-3, Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient
Stroke recurrence at 90 ± 7 days. | 90±7 days post-randomization
  Stroke recurrence
EQ-5D-5L score at 90±7 days | 90±7 days
  The EuroQol 5-Dimension 5-Level Utility Score (EQ-5D-5L utility score) ranges from -0.594 to 1.000 (Chinese value set), assessing health-related quality of life, with higher scores indicating better health status.
Any Intracranial Hemorrhage within 48 hours | Randomization to 48 hours
  Heidelberg Bleeding Classification with clinical worsening criteria.
All-cause mortality at 90 days | 90±7 days post-randomization
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hilkens NA, Casolla B, Leung TW, de Leeuw FE. Stroke. Lancet. 2024 Jun 29;403(10446):2820-2836. doi: 10.1016/S0140-6736(24)00642-1. Epub 2024 May 14. PMID 38759664
- [Background] Powers WJ, Rabinstein AA, Ackerson T, et al (2019) Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for HealthcareProfessionals From the American Heart Association/American Stroke Association. Stroke. https://doi.org/10.1161/STR.0000000000000211
- [Background] Berge E, Whiteley W, Audebert H, De Marchis GM, Fonseca AC, Padiglioni C, de la Ossa NP, Strbian D, Tsivgoulis G, Turc G. European Stroke Organisation (ESO) guidelines on intravenous thrombolysis for acute ischaemic stroke. Eur Stroke J. 2021 Mar;6(1):I-LXII. doi: 10.1177/2396987321989865. Epub 2021 Feb 19. PMID 33817340
- [Background] Wang C, Yi X, Zhang B, Liao D, Lin J, Chi L. Clopidogrel plus aspirin prevents early neurologic deterioration and improves 6-month outcome in patients with acute large artery atherosclerosis stroke. Clin Appl Thromb Hemost. 2015 Jul;21(5):453-61. doi: 10.1177/1076029614551823. Epub 2014 Sep 23. PMID 25248816
- [Background] Guo ZN, Zhang KJ, Zhang P, Qu Y, Abuduxukuer R, Nguyen TN, Chen HS, Yang Y. Early tirofiban administration after intravenous thrombolysis in acute ischemic stroke (ADVENT): Study protocol of a multicenter, randomized, double-blind, placebo-controlled clinical trial. Eur Stroke J. 2024 Jun;9(2):510-514. doi: 10.1177/23969873231225069. Epub 2024 Jan 9. PMID 38196129
- [Background] Liu R, Liang Z, Li W, Zhan Y, Xu L, Yang S, Zheng G, Jiang L, Xie L, Sun Z, Hu Y. Adding Tirofiban on Top of Recombinant Tissue Plasminogen Activator May Improve Clinical Outcome in Acute Stroke Patients. J Stroke. 2024 Jan;26(1):121-124. doi: 10.5853/jos.2023.02250. Epub 2024 Jan 30. No abstract available. PMID 38326710
- [Background] Liang Z, Zhang J, Huang S, Yang S, Xu L, Xiang W, Zhang M. Safety and efficacy of low-dose rt-PA with tirofiban to treat acute non-cardiogenic stroke: a single-center randomized controlled study. BMC Neurol. 2022 Jul 27;22(1):280. doi: 10.1186/s12883-022-02808-w. PMID 35897006
- [Background] Yang M, Huo X, Miao Z, Wang Y. Platelet Glycoprotein IIb/IIIa Receptor Inhibitor Tirofiban in Acute Ischemic Stroke. Drugs. 2019 Apr;79(5):515-529. doi: 10.1007/s40265-019-01078-0. PMID 30838514
- [Background] Jiao Y, Wang X, Guan Y, Wang X, Li Z, Xiang X, Zhang Z. Therapeutic Efficacy of Tirofiban Combined With Thrombus Aspiration and Stent Thrombectomy in the Treatment of Large Vessel Occlusion Ischemic Stroke. Neurologist. 2025 May 1;30(3):140-144. doi: 10.1097/NRL.0000000000000603. PMID 39648705
- [Background] Zhang Y, Zhang QQ, Fu C, Wang L, Zhang GQ, Cao PW, Chen GF, Fu XM. Clinical efficacy of tirofiban combined with a Solitaire stent in treating acute ischemic stroke. Braz J Med Biol Res. 2019;52(10):e8396. doi: 10.1590/1414-431X20198396. Epub 2019 Sep 16. PMID 31531525
- [Background] Higgins JPT, Thomas J, Chandler J, et al (editors). Cochrane Handbook for Systematic Reviews of Interventions version 6.4 (updated August 2023). Cochrane, 2023. Available from www.training.cochrane.org/handbook.
- [Background] de Almeida Monteiro G, Leite M, Goncalves OR, Ferreira MY, Mutarelli A, Marinheiro G, Araujo B, Leal PRL, Ribeiro EML, Figueiredo EG, Telles JPM. Efficacy and safety of intravenous tirofiban combined with reperfusion therapy versus reperfusion therapy alone in acute ischemic stroke: a meta-analysis of randomized controlled trials. J Thromb Thrombolysis. 2025 Apr;58(4):526-537. doi: 10.1007/s11239-025-03094-2. Epub 2025 Apr 1. PMID 40167884